CLINICAL TRIAL: NCT05458687
Title: Traditional Chinese Medicine for Complications in Critically Ill Patients: a Randomized Control Trial
Brief Title: Traditional Chinese Medicine for Complications in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH111-REC3-064
Record Dates: First submitted 2022-06-28; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Critically Ill Patients
Keywords: Traditional Chinese Medicine, intensive care,
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): * Chinese herbal medicine decoction.
  * Acupuncture or Laser acupuncture pen treatment.
  * Acupoint Tuina massage.
  * Acupoint application of traditional Chinese herbal medicinal cake.
  * Nursing and health education and guidance.
  * Diet and health education.
  Interventions: Other: Chinese herbal medicine decoction、Acupuncture or Laser acupuncture pen treatment、Acupoint Tuina massage、Acupoint application、Nursing/Diet and health education and guidance
- control group (No Intervention): * Nursing and health education and guidance
  * Diet and health education

INTERVENTIONS:
Other: Chinese herbal medicine decoction、Acupuncture or Laser acupuncture pen treatment、Acupoint Tuina massage、Acupoint application、Nursing/Diet and health education and guidance — * Chinese herbal medicine decoction: prescribed three times a day, seven days a week, and lasts for up to one weeks.
  * Acupuncture or Laser acupuncture pen treatment: twice a week, once for 20 minutes,up to a total of one week.
  * Acupoint Tuina massage: once a day for up to 20 minutes each time, for up to a week.
  * Acupoint application of traditional Chinese herbal medicinal cake: Apply warm navel ointment in our hospital to CV 4 (Guanyuan) point every day, and remove after getting up the next day, seven days a week for up to one week.
  * Nursing and health education and guidance: teach the patients and their family members the matters needing attention in daily life.
  * Diet and health education:give personalized Traditional Chinese Medicine diet guidance and recommendations in accordance with Traditional Chinese Medicine physique syndrome.
  Arms: intervention group

SUMMARY:
The purpose of this study was to examine the impact of Chinese medicine on common problems in intensive care units.

DETAILED DESCRIPTION:
Introduction: Intensive care unit is a special department in the health care facility. Although with highly development of modern medicine nowadays, the average mortality rate in Intensive care unit is still around 7 to 20 %. There are a few tricky problems that intensivists and intensive care nurses faced very often, including intensive care unit delirium, arrythmia and poor digestion problem that will all affect the mortality and morbidity rate of critical care patients. Traditional Chinese Medicine can possibly provide a series of interventions that can alleviate those conditions.

Methods: A randomized control trial will examine the effect of traditional Chinese Medicine interventions vs. routine intensive care unit care. The patients will be randomly divided 1:1 into one of two groups. A total of 80 intensive care patient will have to meet the following criteria: age 20-90, two or less inotropic medicine use. Interventions such as: Chinese herbal medicine decoction, acupuncture, laser acupuncture, Chinese Tuina massage, herbal medicinal cake applied on acupoint, health education and diet education, will be given based on the patients needs and Traditional Chinese Medicine doctor decision. The main outcomes will be the incidence of arrythmia, delirium, and poor digestion and the severity of pain. The investigators will also record intensive care unit mortality, intensive care unit stays and hospital days.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-90
* newly intensive care unit admission (<48 hours)
* Two or less inotropic medicine prescribed

Exclusion Criteria:

* Clinically unstable: receiving more than inotropic agents.
* Coagulopathy: Prolong Prothrombin Time、activated Partial Thromboplastin Time more than 4 times

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
The main outcomes will be the incidence of arrhythmia, delirium, and poor digestion and the severity of pain. | ICDSC、RASS、BPS record by everyday.
  For delirium use the Intensive Care Delirium Screening Checklist (ICDSC) score of:0~8.
  And Richmond Agitation-Sedation Scale (RASS) score of: -5~+4. For pain use the Behavioral pain scale(BPS) score of:3~12.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan